CLINICAL TRIAL: NCT07018570
Title: An Open Label Phase 2 Study of Total Neoadjuvant Therapy (TNT) Consisting of FLOT With Pembrolizumab and Short Radiation for Patients With Locally Advanced Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kohei Shitara, Chief of Gastroenterology and Gastrointestinal Oncology Division, National Cancer Center Hospital East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC2301
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: Gastroesophageal Junction (GEJ) Adenocarcinoma
Keywords: Esophagogastric junction carcinoma; Total neoadjuvant therapy; TNT; Radiation; Surgery; Pembrolizumab; FLOT; Chemotherapy; Non-operative management; QOL; Phase II
MeSH Terms: conditions — Adenocarcinoma | interventions — pembrolizumab; Docetaxel; Oxaliplatin; Leucovorin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab plus FLOT, Ratiation (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Docetaxel; Drug: Oxaliplatin; Drug: Levofolinate; Drug: Fluorouracil (5-FU); Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg will be administered via intravenous infusion over 30 minutes, twice at 21-day intervals.
Drug: Docetaxel — Docetaxel 50 mg/m2 will be administered over 60 minutes.
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2 will be administered over 2 hours.
Drug: Levofolinate — Leucovorin 200 mg/m2 will be administered over 2 hours.
Drug: Fluorouracil (5-FU) — 5-FU 2600 mg/m2 will be administered over 24 hours.
Radiation: Radiation Therapy — 25Gy (5Gy×5fr)

SUMMARY:
This study is to evaluate the effectiveness of treatment for esophagogastric junction carcinoma, total neoadjuvant therapy (TNT) including pembrolizumab and FLOT is conducted, aiming to choose between surgery or organ preservation treatment strategies.

DETAILED DESCRIPTION:
In Immunochemotherapy before short-term radiation therapy, pembrolizumab 200mg will be intravenously infused at 21-day intervals for 2 doses. FLOT (docetaxel 50 mg/m2, oxaliplatin 85 mg/m2, leucovorin 200mg/m2, 5-FU 2600 mg/m2) will be intravenously infused at 14-day intervals for 2 doses.

Regarding short-term radiotherapy, irradiation will be delivered from day1 to day5, with a dose of 5 Gy per fraction for a total of 25 Gy.

In Immunochemotherapy after short-term radiation therapy, pembrolizumab 200mg will be intravenously infused on day 8. FLOT will be intravenously infused on day 1 and day15.

If CR or Near CR is achieved after the first and second efficacy assessment, pembrolizumab 200mg will be intravenously infused at 21-day intervals for 14 doses and FLOT will be intravenously infused at 14-day intervals for 4 doses as immunochemotherapy as non-operative management (NOM).

If CR or Near CR is not achieved after the first or second efficacy assessment, surgery will be performed. And then pembrolizumab 200mg will be intravenously infused at 21-day intervals for 14 doses and FLOT will be intravenously infused at 14-day intervals for 4 doses as Postoperative adjuvant immunochemotherapy.

ELIGIBILITY:
<Inclusion Criteria>

1. Patients with histologically confirmed esophagogastric junction adenocarcinoma.
2. Patients who are naive to systemic therapy and have esophagogastric junction carcinoma of Siewert Type I to III classified as T: 2-4, N: any, and M: 0 according to the 8th edition of the UICC-TNM classification.
3. Patients aged 18 years or older as of the day of informed consent.
4. Patients with ECOG Performance Status (PS) 0 or 1.
5. Patients whose most recent laboratory values within 14 days before registration meet all of the following criteria (testing on the same day of the week two weeks before the date of registration is acceptable).

[1] Neutrophil count ≥1,500/mm3 [2] Hemoglobin ≥9.0 g/dL [3] Platelet counts ≥100,000/mm3 [4] Total bilirubin ≤1.5 mg/dL [5] AST (GOT) ≤100 IU/L [6] ALT (GPT) ≤100 IU/L [7] Serum creatinine ≤1.5 mg/dL 6) Patients who did not receive blood transfusion within 7 days before registration (ineligible if transfusion was performed on the same day of the week one week before the date of registration).

7)Female patients of childbearing potential who tested negative for pregnancy within 14 days before registration. Male and female patients who have agreed to practice appropriate highly effective contraception with low user dependency during the study and for up to 120 days after discontinuation of the investigational drug.

8)Patients who have given consent to provide samples for biomarker analysis. 9)Patients who have given their own written consent to participate in the study

<Exclusion Criteria>

1. Patients with a history of using an anti-PD-1, anti-PD-L1, or anti-PD-L2 antibody.
2. Patients with a history of acute coronary syndrome (including myocardial infarction and angina unstable), coronary angioplasty, or stent implantation within 6 months before registration.
3. Patients with a history or findings of congestive heart failure of Class II or higher according to the New York Heart Association (NYHA) classification of cardiac function.
4. Patient with active double cancers [simultaneous double cancers and metachronous double cancers with a disease-free interval of ≤2 years. However, carcinoma in situ or lesions equivalent to intramucosal carcinoma judged to have been cured by local treatment shall not be included in active double cancers].
5. Patients with serious (requiring hospitalization) complications (e.g., intestinal paralysis, intestinal obstruction, pulmonary fibrosis, difficult-to-control diabetes mellitus, cardiac failure, myocardial infarction, angina unstable, renal failure, hepatic failure, psychiatric disorder, cerebrovascular disorder).
6. Patients with active hepatitis B (HBs antigen positive) or hepatitis C.
7. Patients with a history of HIV.
8. Patients with complicated interstitial lung disease/pneumonitis or with a history of (non-infectious) interstitial lung disease/pneumonitis requiring steroid administration.
9. Patients who received a live vaccine within 30 days before the start of investigational drug administration.
10. Patients with concomitant autoimmune disease or a history of chronic or recurrent autoimmune disease.
11. Patients who require systemic corticosteroids (except for prophylactic administration for testing or allergic reactions, or temporary use to reduce edema associated with radiotherapy) or immunosuppressive medication, or those who have received any of these treatments within 14 days before registration in this study.
12. Patients with unhealed wounds (requiring sutures, antimicrobial administration, and cleaning procedures), ulcers, or fractures.
13. Pregnant or lactating patients.
14. Patients who are unwilling or unable to comply with the study protocol.
15. Patients deemed by the investigator to be ineligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
3-year event-free survival (EFS) rate | 3 years

SECONDARY OUTCOMES:
Organ-sparing survival | 3 years
Overall survival (OS) | 3 years
Clinical response rate | 3 years
Clinical complete response rate | 3 years
Major pathological response rate (MPR rate) | 3 years
Pathological complete response rate (pCR rate) | 3 years
R0 resection rate (R0 rate) | 3 years
TNT completion rate | 3 years
Treatment completion rate | 3 years
Adverse event incidence rate | 3 years
Post-treatment ctDNA clearance | 3 years
EORTC QLQ-C30 | 3 years
  We are reporting scores from the EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30).
  The scores were transformed to a 0-100 scale following the official EORTC scoring manual. For functional scales and global health status, higher scores indicate a better outcome. For symptom scales/items, higher scores indicate a worse outcome.
EORTC QLQ-OG25 | 3 years
  We are reporting scores from the EORTC QLQ-OG25 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Oesophago-Gastric module).
  The scores were transformed to a 0-100 scale following the official EORTC scoring manual. All scales and single items in the QLQ-OG25 are symptom-based. Therefore, higher scores indicate worse symptoms or poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan

IPD SHARING:
Plan to Share IPD: No